CLINICAL TRIAL: NCT01790646
Title: Learning and Performance of Glidescope® Videolaryngoscope Intubation in Anesthesiologists Trained in Direct Laryngoscopy: a "in Vivo" Study
Brief Title: Learning and Performance of Glidescope® Videolaryngoscope Intubation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Massimo Lamperti, Vice-project coordinator, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Other Study IDs: INCCB 2012-02
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Anesthesia Intubation Complication
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients undergoing general anesthesia: every elective patient undergoing general anesthesia for neurosurgical procedures with endotracheal intubation
  Interventions: Other: intubation

INTERVENTIONS:
Other: intubation — intubation using Glidescope videolaryngoscope

SUMMARY:
Glidescope laryngoscope was introduced as a novel tool for difficult intubation. Its learning curve was prooved on manikin but not in adult patients.

DETAILED DESCRIPTION:
Glidescope® Videolaryngoscope is an angulated rigid optical device introduced in clinical practice in 2004 to facilitate endotracheal intubation.

Since its introduction potential benefits of this instrument might lie with use in patients with clinical features indicating difficult laryngoscopy or it being used as a rescue method following failed direct laryngoscopy. In a few centers was proposed and used routinely.

The performance of Glidescope® was studied in easy and difficult scenarios, in vivo and on manikins and compared with the reference standard McIntosh direct laryngoscopy. In patients with predicted or simulated difficult intubation, despite glottis visualization was improved with Glidescope®, the introduction of the tube in trachea was difficult the same as with McIntosh laryngoscopy. Training of operators before to entertain the trials varied from 20 to 50 Glidescope successful intubations. In an observational study Aziz et al. demonstrated in the two Institutions involved that the GlideScope® was used more frequently at the Institution were the failure rate was significantly lower. At this , 51 providers performed mean 21.7 GlideScope® intubations while at the other 91 providers performed 9.9 intubations.

These data highlight the important issue of how many Glidescope® intubations a provider should complete to reach a definitive clinical competence in this practice. Until now there is only one study performed on mankin comparing Glidescope® with AirTraq® and McIntosh laryngoscopes in novices . The authors concluded that despite a steep learning curve after 5 intubation difficulties in instrumentation and longer times to intubate persisted with Glidescope® in comparison with the other two devices. Outcome measures were: duration of intubation attempt, modified Cormack grades, dental trauma and difficulty of use.

In vivo both timely insertion of laryngoscope blade and introduction of the tube, no need of help or of external laryngeal displacement should be included to ascertain expertise with this new technology in patients with different grades of difficulty predicted.

ELIGIBILITY:
Inclusion Criteria:

* any patient undergoing GA

Exclusion Criteria:

* patients with predicted difficult intubation undergoing awake intubation

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: elective neurosurgical patients from a tertiary neurosurgical centre
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
number of attempts with Glidescope laryngoscopy necessary for beeing considered proficient | from induction of GA to successful intubation
  from Glidescope blade insertion to succefull introduction of the tracheal tube and tube secured in the trachea with ETCO2 confirmation of tracheal ventilation

SECONDARY OUTCOMES:
Features useful to define a Glidescope intubation successful | successfull intubation
  the following criteria have to be satisfied: one introduction of the laryngoscope, one introduction of the tube, Cormack-leane 1, no external laryngeal displacement, time to intubation <43 seconds, no need for help of an external operator, no complications

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cortellazzi, MD, Principal Investigator — Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Locations (1):
- Istituto Neurologico Besta, Milan, Italy